CLINICAL TRIAL: NCT03700684
Title: A Comparison of Two Forms of Intensive Voice Treatment for Parkinson's Disease
Brief Title: Voice Treatment for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Purdue University (Other)
Responsible Party: Principal Investigator, Kelly Richardson, Associate Professor, University of Massachusetts, Amherst
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-4212; 1R21DC016718-01 (NIH)
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants are stratified by voice severity and assigned to one of three groups: Lee Silverman Voice Treatment (intervention), SpeechVive (intervention), or non-treatment control group (control).
Who Masked: Outcomes Assessor
Masking Description: Data files are coded to mask group assignment, session ID, and testing condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Lee Silverman Voice Treatment (Experimental): Persons with Parkinson's disease receive Lee Silverman Voice Treatment over an eight week period. Four weeks of face-to-face intervention and four weeks of home practice.
  Interventions: Behavioral: Lee Silverman Voice Treatment
- SpeechVive (Experimental): Persons with Parkinson's disease receive eight weeks of voice treatment using the SpeechVive device.
  Interventions: Device: SpeechVive
- Control (Active Comparator): Persons with Parkinsons disease do not receive voice intervention
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Lee Silverman Voice Treatment — Persons with Parkinson's disease receive sixteen hours of voice treatment over a four week period. Participants will practice the vocal exercises at home for an additional four weeks.
  Arms: Lee Silverman Voice Treatment
Device: SpeechVive — Persons with Parkinson's disease wear the SpeechVive device several hours a day over an eight week period during opportunities for communication.
  Arms: SpeechVive
Behavioral: Control — Persons assigned to the non-treatment control group will not participate in voice treatment.
  Arms: Control

SUMMARY:
This study addresses several issues related to the clinical management of speech and voice disorders associated with Parkinson's disease. Two behavioral treatment programs, Lee Silverman Voice Treatment and SpeechVive, are assessed in their ability to improve communication in persons with Parkinson's disease.

DETAILED DESCRIPTION:
Surgical and pharmacological management of the motor-based symptoms of PD has made great strides over the last few decades. The behavioral management of the speech and voice symptoms however, has not grown by the same leaps and bounds. Despite the prevalence of speech and voice symptoms associated with PD, few evidence-based treatment options are currently available. In the face of good efficacy data, the Lee Silverman Voice Treatment (LSVT LOUD) program continues to be the gold standard for voice treatment. LSVT LOUD trains patients to monitor and adjust their vocal intensity when they perceive that their voice is soft. Therefore, the success of LSVT LOUD is predicated, in part, on an individual's ability to self-monitor and self-cue (internal cueing) during speech production. While LSVT LOUD has fostered significant improvements in communication for many patients with PD, not all patients respond to treatment. It has been postulated that underlying sensory and cognitive factors may hinder treatment outcomes. A new behavioral treatment for speech and voice impairment has recently been introduced. The SpeechVive, a small in-the-ear device, uses an external noise cue to elicit louder speech. While LSVT LOUD and the SpeechVive have both been shown to significantly increase sound pressure level (SPL) in patients with PD, the physiologic adjustments supporting these changes in SPL remain unclear. This is an important area of study for two reasons. First, both treatments are exercised-based programs, yet the physiologic changes associated with these treatments are not well understood. Second, there is evidence to suggest that the use of an external cue, such as the noise cue used in SpeechVive training, elicits more efficient respiratory patterns in neurologically-healthy and neurologically-involved patients, in comparison to self-initiated cueing strategies, such as those used in LSVT LOUD. This study proposes to compare the influence of cueing strategy on treatment outcomes by examining simultaneous respiratory-laryngeal adjustments before and after participation in LSVT LOUD (internal cueing) and SpeechVive (external cueing) training. It is important to study respiratory-laryngeal interactions because both of these subsystems contribute to vocal intensity regulation. In addition, exercise physiology studies have indicated that internal and external forms of cueing elicit different perceptions of physical and mental effort during exercise. It is important to understand the patients' level of perceived physical and mental effort, associated with each treatment program, as these variables can effect adherence to the treatment regime. In summary, the proposed study is intended to 1) fill a critical void in the investigator's understanding of respiratory-laryngeal adjustments used to support increased SPL under two evidence-based behavioral voice treatment programs, and 2) to better understand how patients' perceptions of physical and mental effort are shaped by each treatment paradigm. The information generated in this study could potentially lead to more efficient voice rehabilitation for persons with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease
* Problems with speech loudness due to Parkinson's disease
* No asthma or other respiratory problems
* No head, neck or chest surgery (Pacemaker surgery is okay)
* Non-smoking for the last 5 years
* Not currently participating in another treatment study
* Typical cognitive skills
* Free of symptoms of depression
* Unaided hearing in at least one ear
* No voice therapy or voice therapy maintenance within the last 12 months

Exclusion Criteria:

* Other neurological diseases, other than Parkinson's disease
* History of asthma or respiratory problems
* Head, neck or chest surgery
* Smoker within the last 5 years
* Currently involved in another treatment study
* Decreased cognition
* Symptoms of depression
* Wear a hearing aid in both ears
* Participated in voice therapy within the last 12 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Richardson, Ph.D., Principal Investigator — University of Massachusetts, Amherst
Locations (2):
- United States (2):
  - Purdue University, West Lafayette, Indiana
  - University of Massachusetts Amherst, Amherst, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The data from the persons with Parkinson's disease will include perceptions of physical and mental effort, objective measures of speech, voice, and respiratory function.
Time Frame: Data will become available once it has been deidentified and published in peer-reviewed journals.
Access Criteria: Any researcher requesting access to these data will need to submit to Kelly Richardson the following:
  1. Name and institution of PI
  2. Proof of institutional appointment
  3. Names and roles for all individuals who will access the data for the planned analysis
  4. Detailed plan for the use of the data
  5. Timeline for the use and publication of the analysis.

REFERENCES:
- [Result] Stathopoulos ET, Huber JE, Richardson K, Kamphaus J, DeCicco D, Darling M, Fulcher K, Sussman JE. Increased vocal intensity due to the Lombard effect in speakers with Parkinson's disease: simultaneous laryngeal and respiratory strategies. J Commun Disord. 2014 Mar-Apr;48:1-17. doi: 10.1016/j.jcomdis.2013.12.001. Epub 2013 Dec 28. PMID 24438910
- [Result] Richardson K, Sussman JE, Stathopoulos ET. The effect of increased vocal intensity on interarticulator timing in speakers with Parkinson's disease: a preliminary analysis. J Commun Disord. 2014 Nov-Dec;52:44-64. doi: 10.1016/j.jcomdis.2014.09.004. PMID 25459460
- [Result] Darling M, Huber JE. Changes to articulatory kinematics in response to loudness cues in individuals with Parkinson's disease. J Speech Lang Hear Res. 2011 Oct;54(5):1247-59. doi: 10.1044/1092-4388(2011/10-0024). Epub 2011 Mar 8. PMID 21386044
- [Result] Sadagopan N, Huber JE. Effects of loudness cues on respiration in individuals with Parkinson's disease. Mov Disord. 2007 Apr 15;22(5):651-9. doi: 10.1002/mds.21375. PMID 17266087
- [Result] Huber JE, Darling M. Effect of Parkinson's disease on the production of structured and unstructured speaking tasks: respiratory physiologic and linguistic considerations. J Speech Lang Hear Res. 2011 Feb;54(1):33-46. doi: 10.1044/1092-4388(2010/09-0184). Epub 2010 Sep 15. PMID 20844256

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lee Silverman Voice Treatment | SpeechVive | Control
Started | 12 | 12 | 12
Completed | 12 | 12 | 10
Not Completed | 0 | 0 | 2
Not completed — COVID-19 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lee Silverman Voice Treatment | SpeechVive | Control | Total
Number analyzed (Participants) | 12 | 12 | 10 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (4.88) | 69 (7.52) | 67 (10.7) | 68 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 11
  Male | 9 | 9 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 10 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 12 | 10 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Hoehn & Yahr [Mean (Standard Deviation); unit: Units on a scale] — The Hoehn and Yahr scale is a system used to describe how the symptoms of Parkinson's disease progress. The scale ranges from 1-5 with 1 representing unilateral involvement with minimal or no functional disability and 5 representing confinement to bed or wheelchair unless aided.
  Units on a scale | 2.5 (0.79) | 2.75 (1.05) | 2.60 (1.26) | 2.62 (1.02)

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Changes in Vocal Intensity Will be Assessed Using Acoustic Analysis.
Description: Vocal intensity (dB SPL) will be measured during a reading task and a monologue task. The vocal intensity data reported will be collapsed across the reading and monologue task. Recorded speech samples are captured using a head-mounted microphone. The speech signals are analyzed for vocal intensity using Praat. The pre- to post-treatment change in vocal intensity is reported in decibels. A positive value indicates an increase in vocal intensity post-treatment. A negative value indicates a decrease in vocal intensity post-treatment. We expected to see no change in vocal intensity for the control group as they did not receive voice intervention.
Time Frame: Change from baseline after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | Lee Silverman Voice Treatment | SpeechVive | Control
Number analyzed (Participants) | 12 | 12 | 10
Decibels | 3 (1.4) | 3 (2.5) | 0.26 (0.23)

2. Primary Outcome: Treatment-related Changes in Speech Breathing Will be Assessed Using Respiratory Kinematics.
Description: Changes in speech breathing will be assessed by examining movement in the ribcage and abdominal walls (respiratory kinematics) during speech. Non-invasive elasticized bands are fitted around the chest and abdominal walls to monitor movement. Respiratory kinematic measures will be in percentage of vital capacity relative to end-expiratory level. Negative values for lung volume termination indicate that speech was terminated below end-expiratory level. Positive values for lung volume termination indicate that speech was terminated above end-expiratory level. The data reported show the baseline and post-treatment values for lung volume initiation, termination, and excursion as a percentage of vital capacity relative to end-expiratory level.
Time Frame: Change from baseline after 8 weeks of treatment
Population: The primary goal was to ascertain the impact of internal cueing (SpeechVive) and external cueing (Lee Silverman Voice Treatment) on respiratory mechanics. To achieve this goal, and to ensure adequate statistical power was maintained, a direct treatment group comparison was undertaken. As a result, the clinical controls, who did not receive any form of intervention, were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: percent change in vital capacity
Arm/Group | Lee Silverman Voice Treatment | SpeechVive
Number analyzed (Participants) | 12 | 12
percent change in vital capacity
  Lung volume initiation (baseline) | 22.89 (20.14) | 21.75 (13.31)
  Lung volume initiation (post-treatment) | 17.87 (15.81) | 20.73 (8.90)
  Lung volume termination (baseline) | 5.84 (16.95) | 6.41 (11.78)
  Lung volume termination (post-treatment) | -6.37 (16.75) | 5.37 (7.90)
  Lung volume excursion (baseline) | 17.05 (12.79) | 15.34 (10.21)
  Lung volume excursion (post-treatment) | 24.24 (17.60) | 15.36 (9.68)

3. Primary Outcome: Treatment-related Changes in Speech Breathing Will be Assessed Using Laryngeal Aerodynamics (Open Quotient)
Description: Movement of air through the vocal folds will also be assessed during a vowel and sentence production task using a vented mask that fits over the nose and mouth. This allows us to derive estimates of how long the vocal folds are open (open quotient). Pre-treatment and post-treatment values are reported. Open quotient is a unit-less measure.
Time Frame: Change from baseline after 8 weeks of treatment
Population: The primary goal was to ascertain the impact of internal cueing (SpeechVive) and external cueing (Lee Silverman Voice Treatment) on laryngeal aerodynamics. To achieve this goal, and to ensure adequate statistical power was maintained, a direct treatment group comparison was undertaken. As a result, the clinical controls, who did not receive any form of intervention, were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: No unit of measurement
Arm/Group | Lee Silverman Voice Treatment | SpeechVive
Number analyzed (Participants) | 12 | 12
No unit of measurement
  Open Quotient (baseline) | 0.72 (0.05) | 0.71 (0.13)
  Open Quotient (post-treatment) | 0.72 (0.11) | 0.68 (0.12)

4. Primary Outcome: Assessing Mental and Physical Effort Associated With Each Treatment Program Using the Modified National Aeronautics and Space Administration (NASA)-Task Load Index
Description: Ratings of physical and mental effort will be assigned by participants on treatment days using the modified NASA-Task Load Index. Participants rate how much physical effort and mental effort it took to complete treatment each day. Participants will indicate their response using a visual analogue scale (0-100) with the endpoints "no effort" ("0") to "significant effort" ("100"). Data are not reported for the clinical control group as these participants did not receive treatment. Ratings of mental and physical effort are reported separately at baseline and post-treatment.
Time Frame: Change from baseline after 8 weeks of treatment
Population: Controls were excluded as the goal was to ascertain the impact of voice intervention on self-perception of physical and mental effort.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lee Silverman Voice Treatment | SpeechVive
Number analyzed (Participants) | 12 | 12
units on a scale
  Mental effort (baseline) | 60.07 (23.53) | 35.23 (30.19)
  Mental effort (post-treatment) | 67.03 (15.54) | 16.59 (17.70)
  Physical effort (baseline) | 65.32 (18.24) | 22.31 (11.13)
  Physical effort (post-treatment) | 67.59 (20.24) | 10.5 (8.15)

5. Secondary Outcome: Treatment-related Changes in Quality of Life Will be Assessed Using the Parkinson's Disease Questionnaire (PDQ-39)
Description: This 39-item self-report questionnaire is designed to address aspects of functioning and well-being for those affected by Parkinson's disease. The PDQ-39 scores each item on a 5 point scale (0=never, 4=always) and is scored along 8 different scales: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. A summary index score is calculated by averaging the scores across these 8 difference scales. The minimum score is 0 and the maximum score is 100. Lower scores indicate a better quality of life and higher scores indicate a lower quality of life. Summary index scores are reported for baseline and post-treatment.
Time Frame: Change from baseline after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lee Silverman Voice Treatment | SpeechVive | Control
Number analyzed (Participants) | 12 | 12 | 10
score on a scale
  Baseline | 18.61 (10.27) | 23.04 (9.04) | 26.74 (16.95)
  Post-treatment | 18.13 (12.70) | 21.60 (11.32) | 23.95 (16.64)

6. Secondary Outcome: Treatment-related Changes in Communicative Competence Will be Assessed Using the Communicative Participation Item Bank-Short Form Questionnaire
Description: The Communicative Participation Item Bank-Short Form is a 10-item self-report questionnaire that examines how a given condition (e.g. Parkinson's disease) interferes with communication in various situations (e.g. noisy environment). The questionnaire has 10 questions that depict a variety of speaking situations. Each of the 10 questions is assigned a score between 0 (very much) to 3 (not at all). Participants are asked to indicate how much their condition interferes with participation in each situation. The scores are summed to come up with a summary score between 0 and 30. High scores indicate less interference in participation.
Time Frame: Change from baseline after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lee Silverman Voice Treatment | SpeechVive | Control
Number analyzed (Participants) | 12 | 12 | 10
score on a scale
  Baseline | 19.17 (5.98) | 16.09 (7.99) | 18.3 (4.95)
  Post-treatment | 23 (4.81) | 16.45 (6.12) | 18.78 (8.48)

7. Secondary Outcome: Treatment-related Changes in Activities of Daily Living Assessed by the Voice-related Quality of Life (VR-QOL) Questionnaire
Description: The Voice-related Quality of Life VR-QOL instrument is a 10-item self-report questionnaire that examines the impact of a persons voice impairment on activities of daily living. For each item, participants assign a score between 1 (Not a problem) and 5 (Problem is as bad as can be). A total score is calculated by summing the assigned scores across the 10 items. The minimum total score is 10 and the maximum total score is 50. Higher scores indicate that the voice problem interferes with activities of daily living. The overall VR-QOL score ranges from 10 to 15 (excellent), 16 to 20 (very good), 21 to 25 (good), 26-30 (fair) and scores more than 30 and up to 50 is poor.
Time Frame: Change from baseline after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lee Silverman Voice Treatment | SpeechVive | Control
Number analyzed (Participants) | 12 | 12 | 10
score on a scale
  Baseline | 19 (7.83) | 23.91 (9.09) | 25.1 (6.37)
  Post-treatment | 16.13 (5.19) | 21.27 (5.98) | 21.33 (7.73)

8. Secondary Outcome: Treatment-related Changes in Speech Rate Will be Assessed Using Acoustic Analysis.
Description: While wearing a microphone, participants will read a short passage. The speech samples will be analyzed for speech rate using an acoustic software program. Speech rate is measured and reported in syllables per second. Higher values indicate a faster speech rate and lower values indicate a slower speech rate.
Time Frame: Change from baseline after 8 weeks of treatment
Population: The primary goal was to ascertain the impact of internal cueing (SpeechVive) and external cueing (Lee Silverman Voice Treatment) on speech rate. To achieve this goal, and to ensure adequate statistical power was maintained, a direct treatment group comparison was undertaken. As a result, the clinical controls, who did not receive any form of intervention, were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: Syllables per second
Arm/Group | Lee Silverman Voice Treatment | SpeechVive
Number analyzed (Participants) | 12 | 12
Syllables per second
  Baseline | 3.27 (0.93) | 3.53 (0.86)
  Post-treatment | 3.26 (0.88) | 3.42 (1.02)

9. Secondary Outcome: Treatment-related Changes in Speech Pauses Will be Assessed Using Acoustic Analysis.
Description: While wearing a microphone, participants will read a short passage. These recorded speech samples will be analyzed for the frequency of pauses using an acoustic analysis software program. Pauses are reported as a frequency count (how many occur in a given sample).
Time Frame: Change from baseline after 8 weeks of treatment
Measure: Mean (Standard Deviation); unit: Pauses per sample
Arm/Group | Lee Silverman Voice Treatment | SpeechVive | Control
Number analyzed (Participants) | 12 | 12 | 10
Pauses per sample
  Baseline | 26 (7.65) | 27.19 (14.03) | 26.6 (8.30)
  Post-treatment | 29.88 (6.24) | 27.18 (9.06) | 27.11 (11.99)

10. Primary Outcome: Treatment-related Changes in Speech Breathing Will be Assessed Using Laryngeal Aerodynamics (MFDR)
Description: Movement of air through the vocal folds will also be assessed during a vowel and sentence production task using a vented mask that fits over the nose and mouth. This allows us to derive estimates of how quickly the vocal folds are closing (maximum flow declination rate). Pre-treatment and post-treatment values are reported. Maximum flow declination rate (MFDR) is reported in liters per second per second (L/s/s).
Time Frame: Change from baseline after 8 weeks of treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/s/s
Arm/Group | Lee Silverman Voice Treatment | SpeechVive
Number analyzed (Participants) | 12 | 12
L/s/s
  Maximum flow declination rate (baseline) | 194.31 (83.69) | 239.90 (200.25)
  Maximum flow declination rate (post-treatment) | 179.53 (42.42) | 181.24 (54.73)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: The study protocol involved non-invasive measures and did not put the subject at risk for a serious adverse event.
Arm/Group | Lee Silverman Voice Treatment | SpeechVive | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lee Silverman Voice Treatment (N=12) | SpeechVive (N=12) | Control (N=10)
Balance (General disorders) | 0 (0) | 0 (0) | 1 (1) — Issues with balance and stability may be present in individuals with Parkinson's disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03700684/Prot_SAP_ICF_000.pdf